CLINICAL TRIAL: NCT00090987
Title: A Phase II Trial Of Imatinib Mesylate (Gleevec) In Patients With HIV Related Kaposi's Sarcoma
Brief Title: Imatinib Mesylate in Treating Patients With HIV-Related Kaposi's Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-042; U01CA070019 (NIH); CDR0000380955 (Other: NCI)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Sarcoma
Keywords: AIDS-related Kaposi sarcoma; recurrent Kaposi sarcoma
MeSH Terms: conditions — Sarcoma; AIDS-related Kaposi sarcoma; Sarcoma, Kaposi | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib mesylate (Experimental): Imatinib mesylate (Gleevec) taken 400 mg orally once a day for up to 6 months
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate — 400 mg orally once a day for up to 6 months.
  Other Names: Gleevec

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking the enzymes necessary for their growth.

PURPOSE: This phase II trial is studying how well imatinib mesylate works in treating patients with HIV-related Kaposi's sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine clinical response in patients with HIV-related Kaposi's sarcoma treated with imatinib mesylate.

Secondary

* Determine the inhibition of platelet-derived growth factor receptors, as determined by immunohistochemistry, in patients treated with this drug.
* Determine cytokine profiles before and after treatment with this drug in these patients.
* Determine the pharmacokinetic profile of this drug and antiretrovirals in these patients.
* Determine mechanisms of primary and secondary resistance to this drug in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral imatinib mesylate once daily. Treatment continues for up to 1 year in the absence of disease progression or unacceptable toxicity.

Patients are followed at 30 days.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Kaposi's sarcoma (KS) involving at least 1 of the following areas:

  * Skin
  * Lymph nodes
  * Oral cavity
  * Gastrointestinal tract*
  * Lungs* NOTE: *Must be asymptomatic or minimally symptomatic AND does not require systemic cytotoxic therapy
* Serological documentation of HIV infection, as evidenced by positive enzyme-linked immunosorbent assay (ELISA), Western Blot test, or other federally approved licensed HIV test
* At least 5 measurable, non-irradiated, cutaneous indicator lesions

  * Patients must have 3 lesions at least 5 x 5 mm that are accessible for 4 mm punch biopsy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* At least 3 months

Hematopoietic

* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 75,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal

  * Patients with elevated bilirubin secondary to indinavir or atazanavir allowed provided total bilirubin is < 3.5 mg/dL AND direct bilirubin is normal
* No acute or known chronic liver disease (e.g., chronic active hepatitis or cirrhosis)

  * Hepatitis C infection with minimal or no fibrosis on liver biopsy allowed

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 60 mL/min

Cardiovascular

* No New York Heart Association class III or IV cardiac disease
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after study participation
* No concurrent active opportunistic infection
* No other severe and/or life-threatening medical disease
* No other malignancy within the past 5 years except clinically insignificant malignancy not requiring active intervention, basal cell skin cancer, or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior biologic therapy for KS
* More than 2 weeks since prior granulocyte colony-stimulating factor
* No concurrent biologic agents for KS

Chemotherapy

* More than 4 weeks since prior chemotherapy for KS (6 weeks for nitrosoureas or mitomycin)
* No concurrent chemotherapy for KS, including systemic cytotoxic chemotherapy

Endocrine therapy

* No concurrent systemic corticosteroid therapy except replacement doses

Radiotherapy

* See Disease Characteristics
* More than 4 weeks since prior radiotherapy for KS
* No concurrent radiotherapy for KS

Surgery

* More than 2 weeks since prior major surgery

Other

* No prior imatinib mesylate
* More than 60 days since prior local therapy to any KS indicator lesion unless the lesion has progressed since treatment
* More than 4 weeks since prior investigational therapy for KS
* More than 4 weeks since other prior therapy for KS
* More than 14 days since prior acute treatment for an infection or other serious medical illness
* No concurrent warfarin
* No concurrent grapefruit juice
* No other concurrent therapy for KS
* No other concurrent investigational drugs
* Concurrent antiretroviral therapy required except for patients who have exhausted all available treatment options

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Noy, MD, Study Chair — Memorial Sloan Kettering Cancer Center; Henry Koon, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (15):
- United States (15):
  - Moores UCSD Cancer Center, La Jolla, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Floyd & Delores Jones Cancer Institute at Virginia Mason Medical Center, Seattle, Washington

REFERENCES:
- [Background] Berman E, Nicolaides M, Maki RG, Fleisher M, Chanel S, Scheu K, Wilson BA, Heller G, Sauter NP. Altered bone and mineral metabolism in patients receiving imatinib mesylate. N Engl J Med. 2006 May 11;354(19):2006-13. doi: 10.1056/NEJMoa051140. PMID 16687713
- [Background] Kerkela R, Grazette L, Yacobi R, Iliescu C, Patten R, Beahm C, Walters B, Shevtsov S, Pesant S, Clubb FJ, Rosenzweig A, Salomon RN, Van Etten RA, Alroy J, Durand JB, Force T. Cardiotoxicity of the cancer therapeutic agent imatinib mesylate. Nat Med. 2006 Aug;12(8):908-16. doi: 10.1038/nm1446. Epub 2006 Jul 23. PMID 16862153
- [Background] Koon HB, Krown SE, Lee JY, Honda K, Rapisuwon S, Wang Z, Aboulafia D, Reid EG, Rudek MA, Dezube BJ, Noy A. Phase II trial of imatinib in AIDS-associated Kaposi's sarcoma: AIDS Malignancy Consortium Protocol 042. J Clin Oncol. 2014 Feb 10;32(5):402-8. doi: 10.1200/JCO.2012.48.6365. Epub 2013 Dec 30. PMID 24378417

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of Recruitment: August 4, 2005 to August 29, 2007 at 12 AMC clinical centers
Pre-assignment Details: Three patients withdrew from the study before receiving treatment.
Groups:
- Imatinib Mesylate (Gleevec): Imatinib mesylate (Gleevec) is administered 400 mg orally once a day
Period: Overall Study
Arm/Group | Imatinib Mesylate (Gleevec)
Started | 30
Completed | 9
Not Completed | 21
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 7
Not completed — Withdrawal by Subject | 3
Not completed — alternative therapy | 1
Not completed — Non-compliance | 4
Not completed — Incarcerated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Achieve a Clinical Response
Description: Clinical response = Complete Response (absence of residual disease) or Partial Response defined as no new lesions (skin or oral), or no new visceral sites of involvement (or the appearance or worsening of tumor-associated edema or effusions); AND 50% or greater decrease in the number of lesions lasting for >4 weeks; OR Complete flattening of at least 50% of all previously raised lesions OR A 50% decrease in the sum of the products of the largest perpendicular diameters of the marker lesions
Time Frame: 20-24 weeks
Measure: Number; unit: proportion
Arm/Group | Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 30
proportion | 0.33

2. Secondary Outcome: Inhibition of Platelet-derived Growth Factor-receptor as Assessed by Immunohistochemistry
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Cytokine Profiles Before and After Imatinib Therapy
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetic Profile of Imatinib and Antiretrovirals
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Mechanisms of Primary and Secondary Resistance to Imatinib Therapy
Description: Mutations in the juxtamembrane or kinase membrane of the c-kit or PDGF receptors at baseline or time of progression
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Viral Transcription Profile of Kaposi's Sarcoma-associated Herpesvirus
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Imatinib Mesylate (Gleevec)
Serious Adverse Events (participants affected / at risk) | 2/30
Other Adverse Events (participants affected / at risk) | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (Gleevec) (N=30)
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) — Hemorrhage, GI/esophagus
Infection (Infections and infestations) | 1 (1) — Infection with normal ANC or Grade 1-2 Neutrophils of the skin (cellulitis)
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Imatinib Mesylate (Gleevec) (N=30)
ALT, SGPT (Metabolism and nutrition disorders) | 2 (2)
Alkaline Phosphatase (Metabolism and nutrition disorders) | 3 (3)
Amylase (Metabolism and nutrition disorders) | 3 (10)
Anorexia (Gastrointestinal disorders) | 3 (3)
Blood/Bone Marrow (Blood and lymphatic system disorders) | 2 (3)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
CPK (Metabolism and nutrition disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Dermatology/skin, other (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 6 (7)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema, limb (Blood and lymphatic system disorders) | 6 (8)
Fatigue (General disorders) | 5 (8)
Gastrointestinal, other (Gastrointestinal disorders) | 2 (2)
Hemoglobin (Blood and lymphatic system disorders) | 6 (7)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 5 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (9)
Insomnia (General disorders) | 2 (2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 4 (6)
Metabolic/laboratory other (Metabolism and nutrition disorders) | 3 (4)
Nausea (Gastrointestinal disorders) | 10 (14)
Neutrophil Count (Blood and lymphatic system disorders) | 4 (7)
Pain, abdominal (Gastrointestinal disorders) | 2 (2)
Pain, back (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, chest (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pain, extremity (Musculoskeletal and connective tissue disorders) | 6 (6)
Pain, muscle (Musculoskeletal and connective tissue disorders) | 3 (4)
Platelets (Blood and lymphatic system disorders) | 2 (2)
Taste Alteration (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (9)
Abdominal bloating (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2007-07-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT00090987/Prot_SAP_001.pdf